CLINICAL TRIAL: NCT01251224
Title: Mouse Allergen and Asthma Intervention Trial
Acronym: MAAIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Children's Hospital (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Elizabeth Matsui, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01AI083238 (NIH)
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Mouse Allergy; Mouse Allergen Exposure
Keywords: asthma; mouse allergen; environmental intervention
MeSH Terms: conditions — Asthma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Group (Active Comparator): This group will receive IPM education at baseline, and then the full IPM intervention after completing the study.
  Interventions: Other: Education
- IPM Group (Experimental): This group will receive the full IPM intervention at baseline.
  Interventions: Other: Integrated Pest Management

INTERVENTIONS:
Other: Integrated Pest Management — The IPM intervention will include professional mouse abatement, two HEPA filters, targeted cleaning, education about IPM, and allergen-proof mattress and pillow encasements. The intervention will be delivered at baseline to the IPM Group, and then repeated if recurrent or persistent mouse infestation is present.
  Arms: IPM Group
Other: Education — This group will receive education about mouse IPM.
  Arms: Education Group

SUMMARY:
The MAAIT is a randomized, controlled trial of a home intervention to reduce mouse allergen exposure in mouse allergic children with asthma and mouse allergen exposure. Participants will be randomized to either the Integrated Pest Management (IPM) Group or the Education Group. The IPM Group will receive professional mouse abatement, education, two HEPA filters, allergen-proof mattress and pillow encasements, and targeted cleaning. The Education Group will receive education about IPM at the beginning of the trial and then after completion of the trial, will receive the IPM intervention. Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* persistent asthma
* exacerbation, previous 12 months
* evidence of mouse sensitization
* high levels of mouse allergen in home
* ages 5-17 years

Exclusion Criteria:

* intermittent asthma
* no exacerbation in previous 12 months
* not sensitized to mouse
* low or undetectable mouse allergen in home
* other lung disease aside from asthma

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2010-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change in asthma symptoms | 0, 3, 6, 9, 12 months
  days of asthma symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's, Boston, Massachusetts

REFERENCES:
- [Derived] Grant T, Phipatanakul W, Perzanowski M, Balcer-Whaley S, Peng RD, Curtin-Brosnan J, Newman M, Cunningham A, Divjan A, Bollinger ME, Wise RA, Matsui EC. Reduction in mouse allergen exposure is associated with greater lung function growth. J Allergy Clin Immunol. 2020 Feb;145(2):646-653.e1. doi: 10.1016/j.jaci.2019.08.043. Epub 2019 Dec 19. PMID 31866099
- [Derived] Ahmed A, Sadreameli SC, Curtin-Brosnan J, Grant T, Phipatanakul W, Perzanowski M, Balcer-Whaley S, Peng R, Newman M, Cunningham A, Divjan A, Bollinger ME, Wise RA, Miller R, Chew G, Matsui EC. Do Baseline Asthma and Allergic Sensitization Characteristics Predict Responsiveness to Mouse Allergen Reduction? J Allergy Clin Immunol Pract. 2020 Feb;8(2):596-602.e3. doi: 10.1016/j.jaip.2019.08.044. Epub 2019 Sep 11. PMID 31520838
- [Derived] Kochis SR, Grant T, Phipatanakul W, Perzanowski M, Balcer-Whaley S, Curtin-Brosnan J, Newman M, Cunningham A, Bollinger ME, Matsui EC. Caregiver-Reported Asthma Control Predicts Future Visits, Independent of Guideline-Based Control Measures. J Allergy Clin Immunol Pract. 2019 May-Jun;7(5):1516-1521.e1. doi: 10.1016/j.jaip.2018.12.030. Epub 2019 Jan 28. PMID 30703536
- [Derived] Matsui EC, Perzanowski M, Peng RD, Wise RA, Balcer-Whaley S, Newman M, Cunningham A, Divjan A, Bollinger ME, Zhai S, Chew G, Miller RL, Phipatanakul W. Effect of an Integrated Pest Management Intervention on Asthma Symptoms Among Mouse-Sensitized Children and Adolescents With Asthma: A Randomized Clinical Trial. JAMA. 2017 Mar 14;317(10):1027-1036. doi: 10.1001/jama.2016.21048. PMID 28264080